CLINICAL TRIAL: NCT00870415
Title: Multicenter (Phase II) Study of Oncoplastic Surgical Techniques for Breast Conservation in Breast Cancers
Brief Title: Breast-Conserving Surgery Techniques in Treating Women With Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Institut du Cancer de Montpellier - Val d'Aurelle (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000633327; CLCC-PHRC-OP-06; CLCC-VA-2006/32; CLCC-ID-RCB-2006-A00694-47; INCA-RECF0638
Record Dates: First submitted 2009-03-26; First posted 2009-03-27 (Estimated); Last update posted 2017-08-21 (Actual); Status verified 2017-08

CONDITIONS: Breast Cancer
Keywords: stage IA breast cancer; stage IB breast cancer; stage II breast cancer; stage IIIA breast cancer; stage IIIC breast cancer; ductal breast carcinoma; invasive ductal breast carcinoma
MeSH Terms: conditions — Breast Neoplasms; Carcinoma, Ductal, Breast

ARMS (1):
- Surgerie (Experimental)
  Interventions: Procedure: quality-of-life assessment; Procedure: therapeutic conventional surgery

INTERVENTIONS:
Procedure: quality-of-life assessment
Procedure: therapeutic conventional surgery

SUMMARY:
RATIONALE: Breast-conserving surgery is a less invasive type of surgery for breast cancer and may have fewer side effects and improve recovery.

PURPOSE: This phase II trial is studying different breast-conserving surgery techniques in treating women with breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Evaluate the percentage of histologically healthy margins maintained during resection in women with breast cancer.

Secondary

* Evaluate local recurrence at 5 years.
* Evaluate aesthetic results.
* Evaluate quality of life using the QLQC30 and BR23 questionnaires.

OUTLINE: This is a multicenter study.

Patients undergo oncoplastic conservative surgery according to defined modalities across the various centers.

Quality of life is assessed periodically.

After completion of study treatment, patients are followed every 6 months for 2 years and then for at least 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Meets 1 of the following criteria:

  * Diagnosis of intraductal breast cancer requiring a wide local resection
  * Diagnosis of infiltrating ductal breast cancer within range
  * Diagnosis of invasive breast cancer that has not responded well to neoadjuvant treatment
* No multicentric tumor
* No gigantomastia
* Hormone receptor status not specified

PATIENT CHARACTERISTICS:

* Menopausal status not specified
* No patients subject to a measure of legal protection or unable to express consent
* No patients deprived of liberty by judicial or administrative decision or hospitalized without patient consent
* Not pregnant or nursing

PRIOR CONCURRENT THERAPY:

* No prior radiotherapy to the diseased breast
* No prior adjuvant treatment
* No concurrent participation in another clinical research study

Ages: 18 Years to 120 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 263 (Actual)
Dates: Start 2007-04; Primary Completion 2009-04 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Percentage of histologically healthy margins maintained during resection | From inclusion to end of intervention

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Rouanet, MD, PhD, Principal Investigator — Institut du Cancer de Montpellier - Val d'Aurelle
Locations (1):
- Centre Regional de Lutte Contre le Cancer - Centre Val d'Aurelle, Montpellier, France